CLINICAL TRIAL: NCT04421703
Title: Scaling up the Med-South Lifestyle Program to Reduce Chronic Disease in Partnership With Rural Communities: Phase 1
Brief Title: Med-South Lifestyle Study: Phase 1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 19-2079
Record Dates: First submitted 2020-05-07; First posted 2020-06-09 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-07

CONDITIONS: Healthy Lifestyle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Distance Collaborative (Experimental): For sites randomized to the distance arm, training will be delivered via web conference, and technical assistance and assessment and feedback will be delivered by phone.
  Interventions: Behavioral: Med-South Lifestyle Program
- Blended in-person/distance collaborative (Experimental): For the QI collaborative arm, training will be delivered in two in-person collaborative meetings; and the remainder of the strategies will be delivered via web-conferencing.
  Interventions: Behavioral: Med-South Lifestyle Program

INTERVENTIONS:
Behavioral: Med-South Lifestyle Program — The Med-South Lifestyle Program is an evidence-based behavior change intervention that translates the PREDIMED (Mediterranean) dietary pattern for a Southeastern US population and includes support for increased physical activity.

SUMMARY:
The purpose of this study is to determine the processes by which a previously proven lifestyle intervention (the Med-South Lifestyle Program) can most effectively and efficiently be translated into public health and clinical practice to positively impact chronic disease risk reduction among mostly minority, rural, and medically underserved populations.

DETAILED DESCRIPTION:
Purpose: Although lifestyle behavior change interventions are widely recommended to improve health, they are not being implemented sufficiently or equitably on a national scale, particularly in rural communities. The research team has developed and tested multiple lifestyle interventions, which have culminated in the Med-South Lifestyle Program (MSLP), an evidence-based behavior change intervention that translates the PREDIMED (Mediterranean) dietary pattern for a Southeastern US population and includes support for increased physical activity. In this research the investigators propose to identify the most effective and efficient way to scale-up the MSLP for use in public health and clinical practices settings so that it reaches minority, rural, and medically underserved populations.

In Phase 1, the investigators will develop, pilot test, and refine implementation strategies that will be used to take the MSLP to scale.

Participants: Phase I participants include up to 80 participants who will receive the MSLP and for whom the study team will collect baseline and follow-up data.

Procedures (methods): An evidence-based framework for scaling-up health interventions will be used to guide Phase I activities. The initial phase involves refining the "scalable unit" which includes the lifestyle program (MSLP), implementation strategies for the sites that will give the program, and strategies UNC will use to train sites on implementing the program. To refine the scalable unit the investigators will apply a descriptive, qualitative design to assess the feasibility and acceptability of the MSLP's intervention and implementation strategies (i.e., what the investigators will scale-up in Phases 2 and 3). In Phase 1, the study team will recruit 2 local health departments and 2 federally qualified health centers as participating sites. Each site will form an implementation team of 2-4 individuals who will go through training on intervention delivery and implementation. Sites will be randomized to receive training either through a distance (webinar) or in-person/collaborative format. Each site will recruit up to 20 participants (for a total of 80 across all sites) to receive the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* English speaking
* Ages 18-80

Exclusion Criteria:

* Malignancy
* Advanced kidney disease (estimated creatinine clearance < 30 mL/min)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Percentage of Eligible Patients Participating | Month 6
  Percentage of each setting's eligible patients who participate in the Med-South Lifestyle Program and the representativeness of participants (age, gender, race/ethnicity) as compared to overall population of eligible patients.
Percentage of Med-South Lifestyle Program Delivered as Intended | Month 6
  To determine delivery fidelity, the study team will measure the degree to which the intervention is delivered as intended as assessed by direct observations and audio file reviews documented by checklist.

SECONDARY OUTCOMES:
Mean Change Number of Fruit and Vegetable Servings Per Day | Baseline, Month 6
  The mean difference in fruit and vegetable servings per day (baseline servings/day - follow-up servings/day) as measured by the Block Fruit-Vegetable-Fiber Screener.
  The Block Fruit-Vegetable-Fiber Screener is a 10-item scale with responses ranging from: (1) Less than 1/week to (5) 2+ a day. Higher scores reflect a better outcome.
Mean Change in Minutes of Physical Activity Per Week | Baseline, Month 6
  Mean difference in minutes of physical activity per week (baseline activity in minutes/week - follow-up activity in minutes/week) as measured by the validated modified RESIDE questionnaire. The RESIDE questionnaire is a 21-item self-administered instrument in which participants recall the frequency, duration, and destination of their walking (for transport and recreation) within and outside of their neighborhood, and cycling activity in a usual week. Higher scores indicate more minutes of activity.
Mean Percent Change in Weight | Baseline, Month 6
  Mean weight change (in kg) from baseline to follow-up expressed as a percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Samuel-Hodge, PhD, Principal Investigator — UNC Chapel Hill; Jennifer Leeman, DrPH, Principal Investigator — UNC Chapel Hill
Locations (3):
- United States (3):
  - Rural Health Group, Norlina, North Carolina
  - Granville-Vance Public Health, Oxford, North Carolina
  - Person Family Medical Center, Roxboro, North Carolina

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samuel-Hodge CD, Gizlice Z, Allgood SD, Bunton AJ, Erskine A, Leeman J, Cykert S. Strengthening community-clinical linkages to reduce cardiovascular disease risk in rural NC: feasibility phase of the CHANGE study. BMC Public Health. 2020 Feb 21;20(1):264. doi: 10.1186/s12889-020-8223-x. PMID 32085707
- [Background] Leeman J, Calancie L, Hartman MA, Escoffery CT, Herrmann AK, Tague LE, Moore AA, Wilson KM, Schreiner M, Samuel-Hodge C. What strategies are used to build practitioners' capacity to implement community-based interventions and are they effective?: a systematic review. Implement Sci. 2015 May 29;10:80. doi: 10.1186/s13012-015-0272-7. PMID 26018220
- [Background] Keyserling TC, Samuel-Hodge CD, Pitts SJ, Garcia BA, Johnston LF, Gizlice Z, Miller CL, Braxton DF, Evenson KR, Smith JC, Davis GB, Quenum EL, Elliott NT, Gross MD, Donahue KE, Halladay JR, Ammerman AS. A community-based lifestyle and weight loss intervention promoting a Mediterranean-style diet pattern evaluated in the stroke belt of North Carolina: the Heart Healthy Lenoir Project. BMC Public Health. 2016 Aug 5;16:732. doi: 10.1186/s12889-016-3370-9. PMID 27495295
- [Background] Cubillos L, Estrada Del Campo Y, Harbi K, Keyserling T, Samuel-Hodge C, Reuland DS. Feasibility and Acceptability of a Clinic-based Mediterranean-style Diet Intervention to Reduce Cardiovascular Risk for Hispanic Americans With Type 2 Diabetes. Diabetes Educ. 2017 Jun;43(3):286-296. doi: 10.1177/0145721717706030. Epub 2017 Apr 21. PMID 28427311
- [Background] Thomas T, Samuel-Hodge CD, Porterfield DS, Alva ML, Leeman J. Scaling Up Diabetes Prevention Programs in North Carolina: Perceptions of Demand From Potential Program Recipients and Providers. Diabetes Educ. 2019 Feb;45(1):116-124. doi: 10.1177/0145721718811564. Epub 2018 Nov 9. No abstract available. PMID 30413136
- [Background] Rohweder C, Wangen M, Black M, Dolinger H, Wolf M, O'Reilly C, Brandt H, Leeman J. Understanding quality improvement collaboratives through an implementation science lens. Prev Med. 2019 Dec;129S:105859. doi: 10.1016/j.ypmed.2019.105859. Epub 2019 Oct 23. PMID 31655174
- [Background] Leeman J, Toles M. What does it take to scale-up a complex intervention? Lessons learned from the Connect-Home transitional care intervention. J Adv Nurs. 2020 Jan;76(1):387-397. doi: 10.1111/jan.14239. Epub 2019 Nov 20. PMID 31642091
- See also: The current study will adapt intervention and dissemination materials from the CHANGE Study. — http://change.web.unc.edu/